CLINICAL TRIAL: NCT04884464
Title: Clinical Evaluation of a Hyaluronic Acid-based Medical Device in Counteracting Aphthous Stomatitis in Adults
Brief Title: Hyaluronic Acid in Counteracting Aphthous Stomatitis
Status: Completed | Type: Observational
Sponsor: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Davide Sisti, PhD, University of Urbino "Carlo Bo"
Other Study IDs: UniUrb_HyalAcid_2021
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Aphthous Stomatitis
Keywords: mucositis; oral ulcers; chlorhexidine; aloe barbadensis; rosa damascena
MeSH Terms: conditions — Stomatitis, Aphthous; Mucositis; Oral Ulcer | interventions — chlorhexidine gluconate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: US Export: No

GROUPS / COHORTS (2):
- Hyaluronic acid-based gel: The composition of the gel, ranked by weight is: xylitol, glycerin, Rosa damascena petal extract, xanthan gum, polycarbophil, hyaluronic acid sodium salt (0.24%), pectin, potassium sorbate, sodium benzoate, panthenol, Aloe barbadensis leaf extract, stevia.
  Interventions: Device: Hyaluronic acid-based gel
- Chlorhexidine gluconate: Chlorhexidine gluconate at a concentration of 0.2%.
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Device: Hyaluronic acid-based gel — Dosage: application of an even coat of 1mm thickness Frequency: 3 times/day (after main meals) Duration: 2 weeks
  Groups: Hyaluronic acid-based gel
Drug: Chlorhexidine Gluconate — Dosage: application of an even coat of 1mm thickness Frequency: 3 times/day (after main meals) Duration: 2 weeks
  Groups: Chlorhexidine gluconate

SUMMARY:
Oral mucosal ulcers can determine a real worsening of the quality of life. Conventional therapy usually lasts not less than 2-3 weeks, and carries a high risk of serious side effects; furthermore, ulcers often recur. The use of hyaluronic acid applied as an adhesive gel over the lesions seems to have potential in terms of efficacy and the avoidance of side effects. Of course, hyaluronic acid-based formulations show different effects and tolerability. In this retrospective observational study, the results obtained using a hyaluronic-acid based medical device applied for 14 days to counteract ulcers in adults will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aphthous stomatitis
* Healthy for other conditions excluding aphthous stomatitis

Exclusion Criteria:

* Taking one of the following in the 45 days prior to the beginning of the study: immunosuppressive, cytotoxic, cortisone, antibiotic, antifungal, hormone therapy (including birth control pills).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects without ethnic limitations, of both sexes and between the ages of 18 and 65, with a diagnosis of aphthous stomatitis, but considered otherwise healthy.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in number of oral lesions | Day 1; Day 3; Day 6; Day 9; Day 12; Day 14
  Change from baseline (Day 1) to Day 14 in the number of oral lesions observed in the two groups
Change in size of oral lesions | Day 1; Day 3; Day 6; Day 9; Day 12; Day 14
  Change from baseline (Day 1) to Day 14 in the size (mm) of oral lesions observed in the two groups

SECONDARY OUTCOMES:
Compliance to treatment | From Day 1 to Day 14
  Number of daily treatments completed, timing of treatment application (hour of the day)
Side effects to treatment | From Day 1 to Day 14
  Dosage Record Treatment Emergent Symptom Scale (DOTES). It uses a Likert scale, going from 1 (no side effects) to 4 (severe side effects).

CONTACTS AND LOCATIONS:
Overall Officials: Davide Sisti, PhD, Principal Investigator — University of Urbino "Carlo Bo"
Locations (1):
- University fo Urbino Carlo Bo, Urbino, Italy

IPD SHARING:
Plan to Share IPD: No